CLINICAL TRIAL: NCT04318301
Title: Hypertension in Patients Hospitalized With COVID-19 in Wuhan, China: A Single-center Retrospective Observational Study
Brief Title: Hypertension in Patients Hospitalized With COVID-19
Acronym: HT-COVID19
Status: Completed | Type: Observational
Sponsor: Zhenhua Zen (Other)
Responsible Party: Sponsor-Investigator, Zhenhua Zen, Associate Professor, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Other Study IDs: HT-COVID19
Record Dates: First submitted 2020-03-20; First posted 2020-03-23 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Hypertension
Keywords: COVID-19; Hypertension; ACE2
MeSH Terms: conditions — COVID-19; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACEI/ARB: COVID-19 patients with hypertension who had previously taken ACEI/ARB for antihypertensive treatment
- non ACEI/ARB: COVID-19 patients with hypertension who had not previously taken ACEI/ARB for antihypertensive treatment

SUMMARY:
Some studies have shown that the main pathogenesis of patients with covid19 is related to ACE2 receptor. Lung is one of the main organs, and there are many ACE2 receptors in cardiovascular system. ACEI / ARB is the main target of antihypertensive drugs. Previous reports suggested that there were large number of patients with covid19 also suffered from hypertension, suggesting that patients with hypertension may be the susceptible to covid19. Therefore, we try to follow up the patients admitted to Hankou hospital to explore the impact of hypertension and hypertension treatment on the severity and prognosis of patients with covid19, so as to provide new methods for the treatment of patients with covid19 in the future.

DETAILED DESCRIPTION:
In December, 2019, a cluster of severe pneumonia cases of unknown cause emerged in Wuhan, China, with clinical presentations greatly resembling viral pneumonia1. Deep sequencing analysis from lower respiratory tract samples indicated a novel coronavirus, which was named 2019 novel coronavirus (2019-nCoV, then named COVID-19). Up to Mar 16, 2020, the total number of patients had risen sharply to 153,546 confirmed cases worldwide (http://2019ncov.chinacdc.cn/2019-nCoV/global.html). The data extracted from 1099 patients with laboratory-confirmed COVID-19 in China from January 29, 2020 showed that hypertension is the most common coexisting illness of COVID-19 patients, ranging from 13.4% in nonsevere patient vs. 23.4% in severe patients, and the total incidence is as high as 15%2. Interestingly, ACE2 is involved in the pathogenesis of both hypertension and SARS-COV-2 pneumonia. The above reasons prompted us to speculate that the organs attacked by SARS-COV-2 might not only be lungs, but also include other ACE2 expression organs, especially cardiovascular system. In addition, patients with comorbid hypertension, especially those with long-term oral ACEI/ARB medication for hypertension, might have different susceptibility and severity levels of pneumonia upon SARS-COV-2 attack. Therefore, we investigated and compared the demographic characteristics, coexisting disease, severity of pneumonia, and the effect of antihypertensive drugs (ACEI/ARB versus non-ACEI/ARB) in patients with COVID-19 coexisting hypertension, thereby, hopefully, to reduce the mortality and morbidity associated with hypertension in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 pneumonia patients diagnosed by WHO criteria

Exclusion Criteria:

* Patients who were younger than 18 years.
* Patients whose entire stay lasted for less than 48 hours.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically confirmed COVID-19 admitted to Hankou Hospital, Wuhan, China from January 5 to March 8, 2020.
Sampling Method: Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2020-03-21 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Rate of Death | From date of admission until the date of death from any cause, up to 60 days
  mortality in 28-day

SECONDARY OUTCOMES:
the severity of pneumonia | From date of admission until the date of discharge or death from any cause, up to 60 days
  evaluate the severity of pneumonia according to CT scans and clinical manifestation

OTHER OUTCOMES:
the length of hospital stay | From date of admission until the date of discharge or death from any cause, up to 60 days
  days from admission to discharge or death

CONTACTS AND LOCATIONS:
Locations (1):
- Hankou Hospital, Hankou, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Li W, Moore MJ, Vasilieva N, Sui J, Wong SK, Berne MA, Somasundaran M, Sullivan JL, Luzuriaga K, Greenough TC, Choe H, Farzan M. Angiotensin-converting enzyme 2 is a functional receptor for the SARS coronavirus. Nature. 2003 Nov 27;426(6965):450-4. doi: 10.1038/nature02145. PMID 14647384
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Wang Z, Chen Z, Zhang L, Wang X, Hao G, Zhang Z, Shao L, Tian Y, Dong Y, Zheng C, Wang J, Zhu M, Weintraub WS, Gao R; China Hypertension Survey Investigators. Status of Hypertension in China: Results From the China Hypertension Survey, 2012-2015. Circulation. 2018 May 29;137(22):2344-2356. doi: 10.1161/CIRCULATIONAHA.117.032380. Epub 2018 Feb 15. PMID 29449338
- [Background] Ferrario CM, Jessup J, Chappell MC, Averill DB, Brosnihan KB, Tallant EA, Diz DI, Gallagher PE. Effect of angiotensin-converting enzyme inhibition and angiotensin II receptor blockers on cardiac angiotensin-converting enzyme 2. Circulation. 2005 May 24;111(20):2605-10. doi: 10.1161/CIRCULATIONAHA.104.510461. Epub 2005 May 16. PMID 15897343
- [Background] Turner AJ, Hiscox JA, Hooper NM. ACE2: from vasopeptidase to SARS virus receptor. Trends Pharmacol Sci. 2004 Jun;25(6):291-4. doi: 10.1016/j.tips.2004.04.001. PMID 15165741
- See also: A Novel Coronavirus From Patients With Pneumonia in China, 2019 — https://pubmed.ncbi.nlm.nih.gov/31978945/?from_single_result=31978945